CLINICAL TRIAL: NCT04855955
Title: Individual Patient Expanded Access Investigation New Drug (IND) Application for Administration of Autologous Human Adipose-Derived Mesenchymal Stem Cells in Alzheimer's Disease
Brief Title: Autologous Human Adipose-Derived Mesenchymal Stem Cells in Alzheimer's Disease
Status: No longer available | Type: Expanded Access
Sponsor: Celltex Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CTXSP0001
Record Dates: First submitted 2021-03-30; First posted 2021-04-22 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer Disease
Keywords: Autologous Adipose-derived Stem Cells (AdMSCs)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Adipose-Derived Mesenchymal Stem Cells

SUMMARY:
This is a single patient emergency expanded access clinical study to assess the safety of administering autologous AdMSCs to an incurable Alzheimer disease patient. The study subject will be evaluated for disease-associated severity according to symptoms, cognitive function, memory, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The patient is diagnosed with later stage of Alzheimer Disease with sever cognitive disability.
* All current anti-Alzheimer medicines cannot prevent disease progression and the patient's mental and physical ability persistently declined
* Patient's legal guardian and caregiver must voluntarily sign an approved written consent form after ample explanation of the proposed therapy.

Exclusion Criteria:

* Current diagnosis of malignancy
* Renal/liver dysfunction: Exceed two times as normal subject
* Pregnant or nursing
* Received other trial drugs within 30 days after participation of this study
* Experienced major surgery or trauma in the last 14 days

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Neel, M.D., Principal Investigator — Little Alsace Urgent Care Center